CLINICAL TRIAL: NCT03724604
Title: A Prospective Cohort Study on NSE/Alb as a Prognostic Biomarker for Lung Cancer Patients in Multicenter
Brief Title: NSE/Alb as a Prognostic Biomarker for Lung Cancer
Acronym: NARPBLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Second Affiliated Hospital of Xi'an Jiaotong University (Other); Shaanxi Provincial Cancer Hospital (Other); Shaanxi Provincial People's Hospital (Other); Xi'an Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2017-020
Record Dates: First submitted 2018-10-28; First posted 2018-10-30 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2018-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Neuron-Specific Enolase; Albumin; Prognostic Biomarker
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high NAR: Neuron-Specific Enolase to Albumin Ratio is higher than 3.2×10-7
  Interventions: Diagnostic Test: Neuron-Specific Enolase to Albumin Ratio
- low NAR: Neuron-Specific Enolase to Albumin Ratio is lower than 3.2×10-7
  Interventions: Diagnostic Test: Neuron-Specific Enolase to Albumin Ratio

INTERVENTIONS:
Diagnostic Test: Neuron-Specific Enolase to Albumin Ratio — Previous studies have shown that inflammation and nutrition-related factors such as CRP/Alb (C-reactive protein-albumin ratio), PLR (platelet-to-lymphocyte ratio), NLR (neutrophil-to-lymphocyte ratio) can help to assess the prognosis of malignant tumors. This study is the first time to combine NSCLC tumor marker NSE and patient nutrition-related indicators Alb to predict the prognosis of patients, trying to find high sensitivity and specificity for NSCLC prognostic indicators to guide clinical work.

SUMMARY:
The incidence and mortality rate of lung cancer is the highest in the world. Current studies have found that tumor markers, inflammatory or nutritional indicators have a good predictive value for the prognosis of patients with non-small cell lung cancer (NSCLC). Neuron specific enolase (NSE) and serum albumin (Alb) are important indicators for monitoring tumor progression and nutritional status in lung cancer patients, respectively. Previous studies suggested that the higher the NSE, the worse prognosis of NSCLC patients, while the lower the Alb, the worse the prognosis of patients with malignant tumors. Through a retrospective study, the investigators found that NAR (NSE Alb Ratio) was higher and prognosis was poorer in patients undergoing NSCLC surgery. This is better than the previous assessment indicators PLR (platelet to lymphocyte ratio), NLR (neutrophil to lymphocyte ratio), AGR (albumin to globulin ratio), NAR can better assess prognosis. Therefore, on the basis of the previous retrospective analysis, the optimal NAR cut-off value was calculated according to ROC curve, and the value was grouped into multi-center prospective cohort study, and the relationship between NAR and other clinical indicators was studied by chi-square test. Univariate and multivariate analysis of Cox proportional hazard regression model was used to determine the prognostic factors. Finally, NSCLC patients were stratified according to tumor stage and pathological classification, and the differences of survival time between high NAR group and low NAR group were compared again under different stages and types, and the different stages of NAR in NSCLC patients were further analyzed. The clinical significance of typing. By exploring and validating the relationship between NAR and the prognosis of NSCLC patients, the investigators try to establish a new prognostic index. Obviously, it has important value for clinical application.

ELIGIBILITY:
Inclusion Criteria:

* (1) pathological diagnosis of non-small cell lung cancer
* (2) 18-70 years of age and no gender restriction.
* (3) patients who were admitted for the first time and underwent routine blood tests, three lung cancer and liver function tests.

Exclusion Criteria:

* (1) pregnant or lactating women
* (2) patients with other malignancies at the same time
* (3) patients with acute and chronic inflammation, autoimmune diseases, and patients with obvious liver and renal insufficiency.
* (4) patients with incomplete clinical and pathological data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample sources: Xi'an Jiaotong University First Affiliated Hospital, Second Affiliated Hospital, Shaanxi Provincial People's Hospital, Shaanxi Provincial Cancer Hospital and other hospitals.
  Subject recruitment process:
  1. Subject screening: Subjects were screened according to inclusion and exclusion criteria.
  2. Recruitment of the research subject: In the course of clinical diagnosis and treatment, the competent doctor recruits.
  3. Subject informed consent: inform patients to collect their clinical data and follow up for clinical studies, signing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years.
  The time from randomization to death due to any cause. The last follow-up time is usually calculated as the time of death for those who have been lost before death.

SECONDARY OUTCOMES:
Disease-free survival | 2 years.
  Refers to the time from randomization to relapse or death due to disease progression. It is usually the end point after radical surgery. DFS is more difficult to record as an end point than OS because it requires careful follow-up and timely detection of disease recurrence. In this study, as an important prognostic indicator for patients undergoing NSCLC surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sida Qin, MD PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First hospital affiliated Xi'an jiaotong university, Xi'an, Shaanxi, China